CLINICAL TRIAL: NCT06956573
Title: Aortic Dimensions in Patients With Fabry Disease
Acronym: DATA-Fab
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Fabien LABOMBARDA, MD, PhD, University Hospital, Caen
Other Study IDs: 5122
Record Dates: First submitted 2025-04-16; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: aorta imaging — Retrospective analysis of imaging data (echocardiography and/or cardiac MRI) in adult patients with Fabry disease to assess ascending aortic diameters.

SUMMARY:
We will conduct a retrospective study aiming to define the characteristics, determinants, and progression of ascending aortic dilatation in adults with Fabry disease, using echocardiography and/or cardiac MRI

ELIGIBILITY:
Inclusion Criteria: a adult patients with genetically confirmed Fabry disease must be able to signed informed consent for participation in the study

Exclusion Criteria:

Patient refusal to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with Fabry disease
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-02 (Estimated); Primary Completion 2025-05-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Maximum ascending aortic diameter measured by transthoracic echocardiography or cardiac MRI, expressed as a Z-score. | At baseline